CLINICAL TRIAL: NCT04769401
Title: Effects of E2 (Estradiol), P4 (Progesterone) and LH Levels on the Day of Transfer and Endometrial Cavity Thickness on Implantation Success in Patients With Frozen-thawed Embryo Transfer Cycle: Prospective Data Analysis
Brief Title: Effects of E2, P4 and LH Levels on the Day of Transfer and Endometrial Cavity Thickness on Implantation Success in Patients With Frozen-thawed Embryo Transfer Cycle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Progesterone study
Record Dates: First submitted 2021-02-14; First posted 2021-02-24 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Infertility; IVF; Progesterone
Keywords: progesterone; infertility; estradiol
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Progesterone group (Experimental): Progesterone level ≥ 10 ng/mL on ET day.
  Interventions: Other: Normal Progesterone group
- Low Progesterone group (Active Comparator): Progesterone level <10 ng/mL on ET day.
  Interventions: Other: Low Progesterone group

INTERVENTIONS:
Other: Normal Progesterone group — Progesteron supplementation was initiated by the use of 100 mg of a vaginal progesterone tablet two times daily (Lutinus, Ferring Pharmaceuticals) plus 250 mg of intramuscular hydroxyprogesterone caproate in oil twice a week (IMHPC) as luteal phase support (referred to as day 0 of progesterone administration).
  Arms: Normal Progesterone group
Other: Low Progesterone group — Progesterone level <10 ng/mL on ET day. If serum progesterone levels were <10 ng/ml at ET day, 25 mg/d of SC progesterone daily (Prolutex) was given to patients and ET was performed on the same day and the blood sample was taken 2 days later to check serum progesterone levels.
  Arms: Low Progesterone group

SUMMARY:
Thanks to recent advances in clinical practice and laboratory, embryo cryopreservation has become the first-line procedure in assisted reproductive technology. Embryo freezing process; Prevention of ovarian hyperstimulation syndrome is becoming an accepted practice for a growing number of indications, including preimplantation genetic testing (PGT), late follicular phase progesterone elevation, and embryo-endometrial asynchrony. Progesterone; plays a key role in the preparation of the endometrial cavity for embryo attachment. Supplementary progesterone preparations can be used to prevent luteal phase defects and provide progesterone support during cycle preparations for frozen-thawed embryo transfer. Our aim in this study is to show the effect of serum progesterone level on pregnancy outcomes on the day of embryo transfer.

DETAILED DESCRIPTION:
This prospective cohort study was conducted at IVF center of Bezmialem University Hospital and Acibadem Health Group between Februrary 2021-September 2021. A total of 234 programmed frozen ultrasound-guided ETs, performed by two physicians (P.O. and C.F.) were included. The study protocol was approved by the Ethical Committee of the Medical Faculty of Bezmialem University. Written informed consent was obtained from all patients. Inclusion criteria were patients underwent IVF between 18 and 41 years old. Exclusion criteria were patients with uncorrected intracavitary structural uterine anomalies including unicornuate, bicornuate or didelphic uterus, recurrent miscarriage, presence of hydrosalpinx, and cycle cancelation. Those undergoing corrective uterine anomalies such as uterine septum, submucosal fibroids, and endometrial polyps were not excluded.

Data collected included age, duration of infertility, type of infertility, indication of IVF, smokers (%),number of previous attempts, serum estradiol (pg/ml), LH (IU/l), progesterone level (ng/ml) and endometrial thickness (mm) prior to progesterone introduction and on embryo transfer day, number of embryos transferred, embryo stage at transfer (Day 3/blastocyst) (%), control progesterone level on post-embryo transfer (ng/ml), the air bubbles (C) at 1 and 60 minutes after embryo transfer,miscarriage, clinical pregnancy rate (the presence of fetal heartbeat visualized by transvaginal ultrasound examination) and ongoing pregnancy rate at 12 weeks of amenorrhea.

Embryo Selection and ET Vitrification on Day 3 or at the blastocyst stage and warming were performed by using commercial vitrification kits according to the manufacturer's instructions. All ETs were performed by two experienced operator (P.O. and C.F.) with Wallace catheter (Smiths Medical International Ltd.) using after-load transfer technique under transabdominal ultrasound guidance with moderately full bladder, without any anesthesia or sedation. The highest quality embryos according to morphology and cleavage criteria were selected for transfer. After the procedure, the patient was kept supine for approximately 60 minutes. Ultrasonography were carried out at 1 and 60 minutes after ET to record the embryo flash position assessed by measuring the distance between the air bubble and the uterine fundus in the coronal image. The embryo flash movement/migration was assessed by measuring the change of the embryo flash position at 60 minutes after ET. When more than one air bubble was seen, the closest one to uterine fundus was used for the measurements. Investigators measured the distance from the lead portion of the air bubble to the uterine fundus.

Endometrial preparation and progesterone support Down-regulation with OCS and a GnRH agonist (Lucrin® 3.75 mg IM, single dose, Ipsen Pharma, Barcelona, Spain) was first done for all patients at the previous cycle and then HRT was used for endometrial preparation at next cycle. Transvaginal ultrasound was performed and serum estradiol, LH and progesterone levels were also measured on the second or third day of menstrual cycle. HRT was started with oral estradiol valerate in a stepwise manner up to 8 mg/day. After 14 days on estrogen supplementation, endometrial thickness was measured by a vaginal 2D ultrasound and serum estradiol, LH and progesterone levels were also measured. If endometrial thickness was >7 mm with a triple layer pattern and quiescent ovaries, serum E2 was >100 pg/ml and the serum P level was <1.5 ng/ml, progesterone supplementation was initiated by the use of 100 mg of a vaginal progesterone tablet two times daily (Lutinus) plus 250 mg of intramuscular hydroxyprogesterone caproate in oil weekly twice as luteal phase support (referred to as day 0 of progesterone administration). Embryo transfer was performed on the day 3 for Day 3 embryos and on day 5 for blastocysts. The blood samples were taken for all patients to measure serum progesterone and estradiol levels at the day of ET. If serum progesterone levels were <10 ng/ml at the day of embryo transfer 25 mg/d of SC progesterone daily (prolutex) were given to patients and a the blood sample was taken 2 days later to check serum progesterone levels. Serum quantitative beta- hCG levels were obtained at 12 days after ET. Progesterone supplementation as luteal phase support was continued at the same dose until 10-12 gestational weeks of viable pregnancies and discontinued if no pregnancy. Oral E2 was discontinued after the presence of fetal heartbeat visualized by transvaginal ultrasound examination.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) ≤25 kg/m2
* between 18 and 41 years old and with FSH levels on cycle day 3 of ≤12 mIU/ml

Exclusion Criteria:

* patients with uncorrected intracavitary structural uterine anomalies including unicornuate, bicornuate or didelphic uterus
* recurrent miscarriage
* presence of hydrosalpinx
* cycle cancelation

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 238 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-11-21 (Actual); Study Completion 2021-11-21 (Actual)

PRIMARY OUTCOMES:
Pregnancy rates | average of 1 year
  Pregnancy rates of the participants

CONTACTS AND LOCATIONS:
Overall Officials: pınar özcan, Principal Investigator — Bezmialem Foundation University
Locations (2):
- Turkey (Türkiye) (2):
  - Acıbadem Kozyatağı Hospital, Istanbul
  - Bezmialem Foundation University, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gardner DK, Lane M. Culture and selection of viable blastocysts: a feasible proposition for human IVF? Hum Reprod Update. 1997 Jul-Aug;3(4):367-82. doi: 10.1093/humupd/3.4.367. PMID 9459282
- [Result] Rienzi L, Gracia C, Maggiulli R, LaBarbera AR, Kaser DJ, Ubaldi FM, Vanderpoel S, Racowsky C. Oocyte, embryo and blastocyst cryopreservation in ART: systematic review and meta-analysis comparing slow-freezing versus vitrification to produce evidence for the development of global guidance. Hum Reprod Update. 2017 Mar 1;23(2):139-155. doi: 10.1093/humupd/dmw038. PMID 27827818
- [Result] Loutradi KE, Kolibianakis EM, Venetis CA, Papanikolaou EG, Pados G, Bontis I, Tarlatzis BC. Cryopreservation of human embryos by vitrification or slow freezing: a systematic review and meta-analysis. Fertil Steril. 2008 Jul;90(1):186-93. doi: 10.1016/j.fertnstert.2007.06.010. Epub 2007 Nov 5. PMID 17980870